CLINICAL TRIAL: NCT02985359
Title: Impact Evaluation of the WFP-Implemented Nutrition Program in Malawi
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United Nations World Food Programme (WFP) (Other); Kamuzu University of Health Sciences (Other); Children's Investment Fund Foundation (Other)
Responsible Party: Principal Investigator, Kristen Hurley, Assistant Professor, Johns Hopkins Bloomberg School of Public Health
Other Study IDs: 00005237
Record Dates: First submitted 2016-06-24; First posted 2016-12-07 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Undernutrition
Keywords: Program impact evaluation; Malawi; Lipid-based nutrient supplements; Social behavior change communication; Childhood stunting
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Collection of Dried Blood Spots
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Comparison district: Existing routine community health services by government
- Program district: In addition to existing routine community health services by the government, daily 20g Nutributter (Lipid-based Nutrient Supplement, LNS) will be provided to children 6 to 24 month of age and caregivers will participate in Social and Behavior Change Communications (SBCC) activities including the promotion of infant and young child feeding (IYCF) behaviors and water, sanitation and hygiene (WASH) behaviors will be conducted with caregivers.
  Interventions: Dietary Supplement: Nutributter; Behavioral: Social Behavioral Change Communication (SBCC)

INTERVENTIONS:
Dietary Supplement: Nutributter — Daily 20g Nutributter provided to children 6 to 24 month of age
  Other Names: Lipid-based nutrient supplement
  Groups: Program district
Behavioral: Social Behavioral Change Communication (SBCC) — Social Behavioral Change Communication (SBCC) activity focused on improving infant and young child feeding (IYCF) practices and water, sanitation, and hygiene (WASH) behaviors through community groups.
  Groups: Program district

SUMMARY:
The goal of this evaluation is to assess the impact of a 3.5 year, World Food Program (WFP) supplemental child feeding and nutrition services program in reducing stunting and improving linear growth in children from 6 through 24 months of age in a rural district of Malawi.

DETAILED DESCRIPTION:
The prevalence of child stunting is high (~47%) in Malawi. In response, the Government of Malawi, with technical support from WFP, launched a 3.5 year of comprehensive nutrition program that provides a small quantity of Lipid-based Nutrient Supplement (LNS) and a comprehensive infant and young child feeding (IYCF) and water and sanitation, and hygiene (WASH) social and behavior change communications (SBCC) package.

The aim of this study is to evaluate the impact of the comprehensive nutrition program in reducing stunting and improving linear growth in children from 6 through 24 months of age and improving infant and young child feeding knowledge and practices in rural Malawi. The study design is quasi-experimental with one program district and one comparison district. The program impact will be evaluated using three rounds of cross-sectional panel data at baseline (January-March, 2014), midline (January-March, 2015), and endline (January-March, 2017). Required sample size for cross-sectional panel is (n = 2400; 1200 per district at each time point) and for pregnant and lactating Women (n = 1200; 600 per district at each time point).

The study also includes the following components:

* Longitudinal study: Two longitudinal cohorts of children (derived from children aged 6-7 months assessed at baseline and mid-line) are followed every 6 months through 24 months of age. Sample size will be ~132; 66 per district in each cohort. As children in the main study, this group will be assessed for their anthropometry.
* Qualitative study: this qualitative study aims to better understand facilitators and barriers to program participation, and factors that influence behavior change among target households. In-depth interviews (IDI) with mothers (n=34) and household members (n=15), and focus group discussions (FGD) with community leaders (n=1 of 11 village chiefs) and program staff (n=1 with 12 community leaders of actions on nutrition (CLAN) and n=2 with a total of 21 care group volunteers [CGV]) will elucidate their perceptions of the program, the Nutributter (NB), and the SBCC messages.
* Process evaluation: The process evaluation will focus on describing and testing the program's implementation theory by evaluating and documenting program inputs, implementation processes and delivery, and outputs. The process evaluation will begin with a broad collection and review of available program documents and data, which are used for the development of the implementation and program theories. To the extent possible, this study will use existing coverage and utilization data from the program's monitoring systems, and will collect additional data needed to fully diagram and understand program implementation activities, procedures, and fidelity to program design. As a final step, the results of the process evaluation will be used to illustrate the program implementation activities that may be expected to contribute to program impacts.
* Cost effectiveness study: In addition to calculating the cost per child covered by the nutrition program in Ntchisi, Malawi, the investigators will use an incremental cost-effectiveness ratio (ICER) approach to report on cost per case of stunting averted and cost per 0.1 unit change in mean length-for-age z-score (LAZ).

ELIGIBILITY:
Inclusion Criteria:

* Children who live in villages sampled for the cross-sectional survey
* Children between 6.0 and 23.9 months of age
* Pregnant and lactating women who live in villages sampled for the cross-sectional survey
* Pregnant or lactating women with a child between the age of 0 to 5.9 months

Exclusion Criteria:

• None

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In both program and comparison sites the investigators will conduct baseline, midline (1 y), and endline (3 y) panel surveys among children 6-23 months of age and pregnant and lactating women in rural Malawi
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2014-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in the prevalence of stunting (%) | Will assess at baseline, midline (1 year), and end line (3 years)
  Children will be measured for their length (cm) among children 6 to 23 months of age. The length measures will be used to create indices of length-for-age (LAZ) z-score based on the WHO child growth standards (WHO Multicentre Growth Reference Study Group 2006). The prevalence of stunting (%) is defined as LAZ<-2. The prevalence of stunting (%) among children 6-23 months of age in the WFP program versus comparison areas at midline (1 year) adjusting for the difference in the prevalence of stunting (%) at baseline between two areas will be a primary outcome at midline (1 year of program implementation). The prevalence of stunting (%) among children 6-23 months of age in the WFP program versus comparison areas at endline (3 years), adjusting for the difference in the prevalence of stunting (%) at baseline between two areas will be a primary outcome at endline (3 years of program implementation).
Change in the prevalence of wasting (%) | Will assess at baseline, midline (1 year), and end line (3 years)
  Children will be measured for their length (cm) and weight (kg) among children 6 to 23 months of age. The length and weight measures will be used to create indices of weight-for-length (WLZ) z-score based on the WHO child growth standards (WHO Multicentre Growth Reference Study Group 2006). The prevalence of wasting (%) is defined as WLZ<-2. The prevalence of wasting (%) among children 6-23 months of age in the WFP program versus comparison areas at midline (1 year) adjusting for the difference in the prevalence of wasting (%) at baseline between two areas will be a primary outcome at midline (1 year of program implementation). The prevalence of wasting (%) among children 6-23 months of age in the WFP program versus comparison areas at endline (3 years), adjusting for the difference in the prevalence of wasting (%) at baseline between two areas will be a primary outcome at endline (3 years of program implementation).
Change in the prevalence of underweight (%) | Will assess at baseline, midline (1 year), and end line (3 years)
  Children will be measured for their weight (kg) among children 6 to 23 months of age. The weight measures will be used to create indices of weight-for-age (WAZ) z-score based on the WHO child growth standards (WHO Multicentre Growth Reference Study Group 2006). The prevalence of underweight (%) is defined as WAZ<-2. The prevalence of underweight (%) among children 6-23 months of age in the WFP program versus comparison areas at midline (1 year) adjusting for the difference in the prevalence of underweight (%) at baseline between two areas will be a primary outcome at midline (1 year of program implementation). The prevalence of underweight (%) among children 6-23 months of age in the WFP program versus comparison areas at endline (3 years), adjusting for the difference in the prevalence of underweight (%) at baseline between two areas will be a primary outcome at endline (3 years of program implementation).

SECONDARY OUTCOMES:
Change in the prevalence of Iron Deficiency Anemia (IDA) (%) | Will assess at baseline and end line (3 years) among a subsample
  Hemoglobin concentration (g/dl) will be assessed on a subsample of mothers and children and used to assess Iron Deficiency Anemia (IDA) (%). The investigators will assess the differences in the IDA (%) among a subsample of mothers and children 6-23 months of age in the WFP program versus comparison areas at endline (3 years), adjusting for the difference in the IDA (%) at baseline between two areas.
Change in the proportion of caregiver knowledge and attitude about infant and young child feeding (IYCF) (%) | Will assess at baseline, midline (1 year), and end line (3 years)
  The investigators will assess the IYCF knowledge and attitude (%) among caregivers of children 6-23 months of age. The proportion of IYCF knowledge and attitude (%) among caregivers in the WFP program versus comparison areas at midline (1 year) adjusting for the difference in the prevalence of IYCF knowledge and attitude (%) at baseline between two areas will be a secondary outcome at midline (1 year of program implementation). The proportion of IYCF knowledge and attitude (%) among caregivers in the WFP program versus comparison areas at endline adjusting for the difference in the prevalence of IYCF knowledge and attitude (%) at baseline between two areas will be a secondary outcome at endline (3 year of program implementation).
Change in the proportion of caregiver knowledge, attitude and practice about infant and young child feeding (IYCF) (%) | Will assess at baseline, midline (1 year), and end line (3 years)
  The investigators will assess the differences in the IYCF knowledge, attitude and practice (%) among caregivers of children 6-23 months of age in the WFP program versus comparison areas at midline (1 year) and at endline (3 years), adjusting for the difference in the IYCF knowledge, attitude, and practice at baseline between two areas.
Change in caregiver practice about handwashing | Will assess at baseline, midline (1 year), and end line (3 years)
  The investigators will assess the hand washing practice (%) among caregivers of children 6-23 months of age. The proportion of hand washing practice (%) among caregivers in the WFP program versus comparison areas at midline (1 year) adjusting for the difference in the prevalence of hand washing practice %) at baseline between two areas will be a secondary outcome at midline (1 year of program implementation). The proportion of hand washing practice (%) among caregivers in the WFP program versus comparison areas at endline adjusting for the difference in the prevalence of hand washing practice (%) at baseline between two areas will be a secondary outcome at endline (3 year of program implementation).

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Hurley, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Wadonda Consult Ltd, Zomba, Malawi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hurley KM, Phuka J, Kang Y, Ruel-Bergeron J, Buckland AJ, Mitra M, Wu L, Klemm RDW, West KP, Christian P. A longitudinal impact evaluation of a comprehensive nutrition program for reducing stunting among children aged 6-23 months in rural Malawi. Am J Clin Nutr. 2021 Jul 1;114(1):248-256. doi: 10.1093/ajcn/nqab010. PMID 33742208
- [Derived] Kang Y, Hurley KM, Ruel-Bergeron J, Monclus AB, Oemcke R, Wu LSF, Mitra M, Phuka J, Klemm R, West KP Jr, Christian P. Household food insecurity is associated with low dietary diversity among pregnant and lactating women in rural Malawi. Public Health Nutr. 2019 Mar;22(4):697-705. doi: 10.1017/S1368980018002719. Epub 2018 Oct 31. PMID 30378520